CLINICAL TRIAL: NCT00485108
Title: Anti-inflammatory Therapy Following Selective Laser Trabeculoplasty (SLT): A Randomized, Masked, Placebo Controlled Study
Brief Title: Anti-inflammatory Therapy Following Selective Laser Trabeculoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Pfizer (Industry); Glaucoma Research Society of Canada (Other)
Responsible Party: Principal Investigator, Dr. Robert Campbell, Assistant Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DJ1
Record Dates: First submitted 2007-06-09; First posted 2007-06-12 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Primary Open Angle Glaucoma; Pseudoexfoliation Glaucoma
Keywords: primary open angle glaucoma; pseudoexfoliation glaucoma; selective laser trabeculoplasty; intra ocular pressure; anti-inflammatory therapy; prednisolone acetate 1%; ketorolac tromethamine 0.5%
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome | interventions — 1(beta)-D-arabinofuranosylcytosine-5'-diphosphate prednisolone; Ketorolac Tromethamine; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Prednisolone 1% eye drop
  Interventions: Drug: prednisolone 1%
- 2 (Active Comparator): ketorolac 0.5% eye drop
  Interventions: Drug: ketorolac 0.5%
- 3 (Placebo Comparator): Artificial Tears (methyl cellulose eye drop)
  Interventions: Drug: Artificial Tears (Methyl cellulose drops)

INTERVENTIONS:
Drug: prednisolone 1% — eye drop once in each eye treated, 4 times / day for 5 days post-laser
  Arms: 1
Drug: ketorolac 0.5% — eye drop once in each eye treated, 4 times / day for 5 days post-laser
  Other Names: Acular
  Arms: 2
Drug: Artificial Tears (Methyl cellulose drops) — eye drop once in each eye treated, 4 times / day for 5 days post-laser
  Other Names: Refresh Tears
  Arms: 3

SUMMARY:
The type of anti-inflammatory medication used post selective laser trabeculoplasty (SLT) may have an impact on the intra-ocular pressure (IOP) lowering effect of SLT. This study will evaluate the IOP lowering effect of SLT following the topical administration of one of the following: prednisolone 1%, ketorolac 0.5% or artificial tears.

DETAILED DESCRIPTION:
Patients who have been chosen to undergo SLT for glaucoma will be randomized to receive one of prednisolone 1%, ketorolac 0.5% or artificial tears four times a day for 5 days following administration of the laser treatment. The IOP will be measured at various time points following SLT: 1 hour, 2 days, 1 week, 1 month, 3 months, 6 months, and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* primary open angle glaucoma, pseudo exfoliation glaucoma

Exclusion Criteria:

* previous incisional glaucoma surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure lowering effect | 1 hour, 2 days, 1 month, 3 months, 6 months and 1 year

SECONDARY OUTCOMES:
intraocular pressure elevation | 1 hour, 2 days, 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Rob J Campbell, MD, MSc, Principal Investigator — Queen's University; Delan Jinapriya, MD, Study Director — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada